CLINICAL TRIAL: NCT01675752
Title: Accuracy of Narrow Band Imaging in Predicting Colonoscopy Surveillance Intervals and Histology of Distal Diminutive Polyps (Small Hyperplastic and Adenomatous Reliability Protocol; SHARP Trial)
Brief Title: Small Hyperplastic and Adenomatous Reliability Protocol
Acronym: SHARP
Status: Completed | Type: Observational
Sponsor: Istituto Clinico Humanitas (Other)
Collaborators: Olympus (Industry)
Responsible Party: Sponsor
Other Study IDs: CE ICH 37/11
Record Dates: First submitted 2012-08-28; First posted 2012-08-30 (Estimated); Last update posted 2012-08-30 (Estimated); Status verified 2012-08

CONDITIONS: Adenomatous Polyp
Keywords: colonoscopy, narrow-band imaging
MeSH Terms: conditions — Adenomatous Polyps

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No

SUMMARY:
1. Protocol Summary Title: SHARP: Small Hyperplastic and Adenomatous Reliability Protocol Purpose: To compare the accuracy of NBI-in vivo differentiation between hyperplastic and adenomatous <10 mm polyps with that of histology in an European multi-center study. To assess variability among endoscopists in NBI accuracy. We also aim to assess whether this technology impacts the appropriateness of surveillance intervals.

Design: 1) Before starting the patient enrollment, the participating endoscopists will attend an internet-based training program on the in vivo differentiation between hyperplastic and adenomatous polyps. Following this course, a qualifying examination will be required for each endoscopist to be included.

2) Patients who are scheduled for screening or diagnostic colonoscopy will be considered for inclusion. Patients with at least one histologically verified <10 mm polyp will be included. In order to measure NBI feasibility, each included polyp will be in vivo assessed by NBI in order to rank between a high- and a low- level of diagnostic confidence, and thereafter will be sent for histological assessment. NBI- and histological accuracy in differentiating between hyperplastic and adenomatous lesions will be analyzed and compared, in order to assess the NBI-sensitivity and specificity. The primary outcomes are to measure the NBI feasibility and accuracy in the study population, and to assess the variability among the endoscopists. Secondary outcome measures will be a cost analysis on how much savings would be achieved by not referring NBI-diagnosed hyperplastic polyps to histology, and a clinical inference on how many patients would be scheduled for an inappropriate post-polypectomy follow up, when follow up schedule is based on NBI classification. Clinical results will be analyzed using various statistical measures of significance.

Clinical Site Locations: 10 European centres with NBI-technology

1 NBI-expert endoscopist for each centre Enrollment: 160 small (<10 mm) polyps at each site Study technology: NBI-Olympus without optical magnification Risk: Non-interventional study.

ELIGIBILITY:
Inclusion Criteria:

* 1. The patient is undergoing colonoscopy for screening, for surveillance in follow-up of previous polypectomy or for diagnostic work-up; 2. The patient is at satisfactory risk to undergo abdominal surgery; 3. The patient must understand and provide written consent for the procedure.

Exclusion Criteria:

* 1. The patient is undergoing colonoscopy for screening, for surveillance in follow-up of previous polypectomy or for diagnostic work-up; 2. The patient is at satisfactory risk to undergo abdominal surgery; 3. The patient must understand and provide written consent for the procedure.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Consecutive adult patients who were referred for elective outpatient colonoscopy will be asked to enroll into this trial if the candidate meets the study inclusion and exclusion criteria.
Sampling Method: Non-Probability Sample
Enrollment: 300 (Actual)
Dates: Start 2011-05; Primary Completion 2012-05 (Actual); Study Completion 2012-07 (Actual)

REFERENCES:
- [Derived] Repici A, Hassan C, Radaelli F, Occhipinti P, De Angelis C, Romeo F, Paggi S, Saettone S, Cisaro F, Spaander M, Sharma P, Kuipers EJ. Accuracy of narrow-band imaging in predicting colonoscopy surveillance intervals and histology of distal diminutive polyps: results from a multicenter, prospective trial. Gastrointest Endosc. 2013 Jul;78(1):106-14. doi: 10.1016/j.gie.2013.01.035. Epub 2013 Apr 11. PMID 23582472